CLINICAL TRIAL: NCT04301596
Title: Assessment of Nutritional Status in Systemic Sclerosis: Prospective Cohort Study in Montpellier University Hospital
Brief Title: Assessment of Nutritional Status in Systemic Sclerosis
Acronym: NUTRISCLER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0409; UF7840 (Other: Montpellier University Hospital)
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SSc patients
  Interventions: Other: Collection of data

INTERVENTIONS:
Other: Collection of data — different set of data will be collected over a 6 months period

SUMMARY:
The main theme of the cohort of systemic sclerosis (SSc) patients is the determination of nutritional status, its evolution and the evaluation of its management in patients with scleroderma.

The main objectives are :

* To determine the incidence of malnutrition and its main determinants (disease characteristics, severity, eating habits, physical activity) in patients with scleroderma.
* For patients with undernutrition at inclusion or at 18 months follow-up:

evaluate the impact of a standardized nutritional intervention (dietary advice, oral supplements, artificial, enteral or parenteral nutrition) on nutritional and disease parameters.

Follow-up visits will take place every 6 months for 2 years. (M6, M12, M18 et M24).

During each visit: a clinical examination, with anthropometric measurements, a 3-day dietary survey and a blood sample (10 ml), completion a multiple-choice of quality of life and physical activity evaluation.

Paraclinical evaluation : echocardiography, lung function tests, screening for osteoporosis (M6 and M18).

If undernutrition is detected during a follow-up visit, the subject will be referred to a specialized service.

ELIGIBILITY:
Inclusion Criteria:

* All SSc patients aged 18 or more
* Patient followed at the Montpellier University Hospital
* Patients must fulfil the American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) 2013 criteria for SSc.
* Health insurance (affiliation to social security)
* Collection of non-opposition to participate in the study

Exclusion Criteria:

* Patient under the protection of justice curatorship / guardianship;
* Patients who have already planned to move out of the region in the next two years, making the follow-up impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients aged 18 or more with scleroderma. From preliminary data obtained in our department, we can estimate that 50% of participants will meet the definition of malnutrition (BMI<21kg/m2 or weigh loss >10% in months) at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2024-10-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of malnutrition | 6 months
  Incidence of malnutrition will be measured as a loss of more than 10% of body weight or a body mass index (BMI) less than 21 kg/m2
Idetification of risk factors associated with malnutrition | 6 months
  Collection of data related to SSc disease burden
Success of the nutritional intervention | 6 months
  body weight gain > 5%

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre MARIA, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No